CLINICAL TRIAL: NCT00420537
Title: Safety and Efficacy of Low-dose Cyclosporine in Association With Everolimus to Minimize Renal Dysfunction in Heart Transplant Recipients
Brief Title: Shift to Everolimus (RAD) Kidney Sparing Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: A cluster of adverse events in everolimus arm was noted.
Sponsor: University of Bologna (Other)
Responsible Party: University of Bologna, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006-003035-78
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-05

CONDITIONS: Kidney Dysfunction; Heart Transplantation
Keywords: Kidney; Heart Transplantation; Creatinine; Glomerular Filtration Rate
MeSH Terms: interventions — Cyclosporine; Mycophenolic Acid; Everolimus

ARMS (2):
- mycophenolate (Active Comparator): Mycophenolate mofetil with cyclosporine trough levels between 100 and 150
  Interventions: Drug: cyclosporine; Drug: Mycophenolate mofetil
- Everolimus (Active Comparator): Everolimus with cyclosporine trough levels between 40 and 90 ng/ml
  Interventions: Drug: cyclosporine; Drug: Everolimus

INTERVENTIONS:
Drug: cyclosporine — cyclosporine trough levels between 100 and 150
  Arms: mycophenolate
Drug: cyclosporine — cyclosporine trough levels between 40 and 90 ng/ml
  Arms: Everolimus
Drug: Mycophenolate mofetil — mycophenolate with low doses
  Arms: mycophenolate
Drug: Everolimus
  Arms: Everolimus

SUMMARY:
The purpose of this study is to verify if the combination of Everolimus with a very low dose of cyclosporine is more effective than the combination of mycophenolate mofetil with low-dose of cyclosporine in reducing the progression of kidney dysfunction in patients with heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Heart Transplant with 1 to 4 years of follow-up
* GFR between 20 and 60 ml/min (calculated with Colkoroft-Gault formula)

Exclusion Criteria:

* Acute rejection in the previous 6 months
* Contraindications to statin therapy
* Ongoing infection
* Ongoing heart failure
* Myocardial infarction or myocardial revascularization after transplant
* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Calculated GFR | One year after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Branzi, MD, Study Chair — Alma Mater Studiorum University of Bologna
Locations (1):
- Policlinico S.Orsola-Malpighi, Bologna, Italy

REFERENCES:
- [Background] Lehmkuhl H, Ross H, Eisen H, Valantine H. Everolimus (certican) in heart transplantation: optimizing renal function through minimizing cyclosporine exposure. Transplant Proc. 2005 Dec;37(10):4145-9. doi: 10.1016/j.transproceed.2005.10.005. PMID 16387066
- [Background] Eisen HJ, Tuzcu EM, Dorent R, Kobashigawa J, Mancini D, Valantine-von Kaeppler HA, Starling RC, Sorensen K, Hummel M, Lind JM, Abeywickrama KH, Bernhardt P; RAD B253 Study Group. Everolimus for the prevention of allograft rejection and vasculopathy in cardiac-transplant recipients. N Engl J Med. 2003 Aug 28;349(9):847-58. doi: 10.1056/NEJMoa022171. PMID 12944570